CLINICAL TRIAL: NCT06232135
Title: Assessment of Reliability of Demirjian Formula for Age Estimation Using Mandibular Third Molar in a Sample of Egyptian Population Using CBT: a Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yara Aladdin Mohamed Shaaban, Master degree student, Cairo University
Other Study IDs: yaraprotocol1893
Record Dates: First submitted 2024-01-20; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Estimated Age Calculated Based on Modified Demirjian Method Using Mandibular Left Third Molar
Keywords: Demirjian; CBCT; age estimation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Females: CBCT scans of the females enrolled in the study are to be analyzed for the assignment of a calcification stage to their lower left third molar according to the modified Demirjian method.
  Interventions: Other: CBCT scan
- Males: CBCT scans of the males enrolled in the study are to be analyzed for the assignment of a calcification stage to their lower left third molar according to the modified Demirjian method.
  Interventions: Other: CBCT scan

INTERVENTIONS:
Other: CBCT scan — analysis of the CBCT scan to assign a calcification stage to the subject's lower left third molar and accordingly calculate the estimated age of each subject

SUMMARY:
Aim: To assess the reliability of age estimation in Egyptian adolescents and young adults using mandibular third molar stages of calcification, based on the Demirjian method, on CBCT scans.

Methodology: 145 CBCT scans for the mandibular left posterior region were collected from the database of the maxillofacial radiology clinic of the faculty of dentistry at Cairo University. The scans were then analyzed using Planmeca Romexis software viewer version 4.6.2.R. The mandibular left 3rd molars were evaluated to determine the calcification stage of each of them based on the modified Demirjian method. According to the assigned calcification stage, the dental age was determined, and then the mean ± SD for each calcification stage was calculated and compared to the chronological age in terms of mean difference and mean absolute error. The correlation between the calculation stage and chronological age was analyzed, and the probability for an individual to be 18 years of age or older in each stage was calculated.

DETAILED DESCRIPTION:
this is a cross-sectional study.

The data collection will be obtained from the database available at the Department of Oral and Maxillofacial Radiology, Faculty of Dentistry, Cairo University. CBCT images will be obtained from Egyptian patients who were referred to the CBCT unit in the oral and maxillofacial radiology departments for different purposes.

* Retrospective Data Analysis will be performed after the CBCT images are pooled from the computer database.
* Exposure parameters of the scans will vary depending on patients' sizes (according to the manufacturer's recommendations).
* Images with 0.4 voxel size or less will be reviewed.
* Evaluation of the calcification of third molar will be done using the reformatted panoramic view of CBCT scans and will be compared with the Demirjian chart (8 stage grading scheme for third molar).
* The third molars from the lower left quadrants will be assessed and categorized into their respective developmental stages given by Demirjian.
* CBCT images will be interpreted by two oral and maxillofacial radiologists (with different experiences) independently; blinded from demographic data of the patients and from the results of each other.
* Each radiologist will evaluate the images for proper determination of the third molar calcification stage and to decide the dental age of the patient according the chart provided by demirjian et al.
* The calcification stage determination will be carried out by one observer and will be repeated later for intra-observer reliability assessment.
* Any disagreement will be solved by consensus between the two observers.
* The chronological age recorded based on his/her date of birth will be correlated with developmental stages of third molar.

The two oral and maxillofacial radiologists interpreting the scans will be blinded from demographic data of the patients and from the results of each other.

A power analysis was designed to have adequate power to apply a statistical test of the null hypothesis that there is no difference would be found between chronological age and developmental age of third molar according to modified Demirjian chart. By adopting an alpha level of (0.05) a beta of (0.2) i.e. power=80% and an effect size (d) of (0.26) calculated based on the results of Mohammed, Rezwana Begum, et al. ; the predicted sample size (n) was a total of (117) cases. Sample size calculation was performed using G*Power version 3.1.9.7 Numerical data will be explored for normality by checking the data distribution, calculating the mean and median values and using Kolmogorov-Smirnov and Shapiro-Wilk tests. If the data was found to be normally distributed, it will be presented as mean and standard deviation values. If the assumption of normality was found to be violated, the data will be presented as median and range values.

Categorical data will be represented as frequency (n) and percentage (%). Categorical data will be represented as frequency (n) and percentage (%) and will be analyzed using chi square test. Numerical data will be explored for normality by checking the data distribution, calculating the mean and median values and using Kolmogorov-Smirnov and Shapiro-Wilk tests. If the data was found to be normally distributed, it will be presented as mean and standard deviation values and Paired t-test will be used for the analysis. If the assumption of normality was found to be violated; the data will be presented as median and range values and will be analyzed using Wilcoxon signed-rank test. The significance level will be set at p ≤0.05 for all tests. Statistical analysis will be performed with IBM® SPSS® Statistics Version 26 for Windows.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian patients with age ranges from 9 to 24 years.
* Complete dental records of radiographs, including the date of birth, date of radiography, and sex.
* Scans showing complete mandibular arch.

Exclusion Criteria:

* Patients below 9 years and above 24 years.
* Any pathology or fractures associated with mandibular third molar.
* Scans with severe metallic artifacts.
* Congenitally absent 3rd molars.

Ages: 9 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — self-representation of gender identity.
Study Population: CBCT scans from the database available at the department of Oral and Maxillofacial Radiology, Faculty of Dentistry, Cairo University.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
accuracy of the modified Demirjian method | 2 weeks
  mean difference between estimated age and chronological age

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry - Cairo university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The age and gender of the participants will be shared. If further information is required, then the invistigator will decide what to share so as not to violate patient privacy.